CLINICAL TRIAL: NCT01320553
Title: Effect of Different Concentrations of SPARC1102 on Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_11_02
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SPARC1102 I (Experimental): 1334H 0.15% eye drops will be administered in both eyes at 3 occasions
  Interventions: Drug: SPARC1102 I
- SPARC1102 II (Experimental): 1334H 0.3% eye drops (solution) will be administered in both eyes at 3 occasions
  Interventions: Drug: SPARC1102 II
- SPARC1102 III (Experimental): 1334H 0.45% eye drops (solution)will be administered in both eyes at 3 occasions
  Interventions: Drug: SPARC1102 III
- Vehicle (Placebo Comparator): Placebo eye drops (solution)will be administered in both eyes at 3 occasions
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SPARC1102 I — SPARC1102 I will be administered in both eyes
  Arms: SPARC1102 I
Drug: SPARC1102 II — SPARC1102 II will be administered in both eyes
  Arms: SPARC1102 II
Drug: SPARC1102 III — SPARC1102 III will be administered in both eyes
  Arms: SPARC1102 III
Drug: Vehicle — Vehicle will be administered in both eyes
  Arms: Vehicle

SUMMARY:
The present study will test if administration of different concentrations of 1334H eyedrops will be effective in treatment of allergic conjunctivitis in people with 10 yrs of age or older.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form and HIPAA document
* Willing and able to comply with all study procedures
* Be at least 10 years of age at the time of enrollment
* LogMar 0.7 or better, in each eye
* History of ocular allergies, and a positive skin and ocular allergic reaction to allergens
* A negative urine pregnancy test if female of childbearing potential and must use adequate birth control throughout the study period

Exclusion Criteria:

* have known contraindications or sensitivities to the use of any of the study medications(s) or their components;
* have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium or a diagnosis of dry eye);
* have a current diagnosis or history of open angle glaucoma or ocular hypertension;
* have had ocular surgical intervention within three (3) months prior to Visit 1 or during the study and/or a history of refractive surgery within the past 6 months;
* have a known history of retinal detachment, diabetic retinopathy, or progressive retinal disease;
* have the presence of an active ocular infection (bacterial, viral or fungal), positive history of an ocular herpetic infection, or preauricular lymphadenopathy at any visit;
* manifest signs or symptoms of clinically active allergic conjunctivitis in either eye at screening or during study
* have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device study within 30 days of the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ORA Inc, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1334 H 0.15%: 1334H 0.15% eye drops will be administered in both eyes at 3 occasions
  1334 H 0.15%: 1334H 0.15% eye drops (solution) will be administered in both eyes at 3 occasions
- 1334 H-0.3%: 1334H 0.3% eye drops (solution) will be administered in both eyes at 3 occasions
  1334 H-0.3%: 1334H 0.3% eye drops (solution) will be administered in both eyes at 3 occasions
- 1334 H-0.45%: 1334H 0.45% eye drops (solution)will be administered in both eyes at 3 occasions
  1334 H-0.45%: 1334H 0.45% eye drops (solution)will be administered in both eyes at 3 occasions
- Vehicle: Vehicle eye drops (solution)will be administered in both eyes at 3 occasions
  Placebo: Placebo eye drops (solution)will be administered in both eyes at 3 occasions
Period: Overall Study
Arm/Group | 1334 H 0.15% | 1334 H-0.3% | 1334 H-0.45% | Vehicle
Started | 31 | 30 | 31 | 30
Completed | 30 | 26 | 29 | 29
Not Completed | 1 | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo eye drops (solution)will be administered in both eyes at 3 occasions
  Placebo: Placebo eye drops (solution)will be administered in both eyes at 3 occasions
- Total: Total of all reporting groups
Arm/Group | 1334 H 0.15% | 1334 H-0.3% | 1334 H-0.45% | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (11.58) | 34.8 (15.42) | 33.7 (15.94) | 40.6 (13.57) | 35.6 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 22 | 21 | 77
  Male | 13 | 14 | 9 | 9 | 45

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular itching evaluated by the subject at 3, 5, and 7 minutes post-challenge (0-4 scale, allowing half unit increments with 0 representing none and 4 representing Incapacitating itch with an irresistible urge to rub) at Visit 5.
Time Frame: Up to 28 days
Population: Of the 122 subjects enrolled in the study, a total of 8 subjects did not complete the study: 1 in the 1334H 0.15% group, 4 in the 1334H 0.3% group, 2 in the 1334H 0.45% group and 1 in the vehicle treated group.
  The Per Protocol population, comprised of all subjects who completed the study with no protocol violations, totaled 107 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1334 H 0.15% | 1334 H-0.3% | 1334 H-0.45% | Vehicle
Number analyzed (Participants) | 29 | 24 | 26 | 28
units on a scale
  7 minutes post challenge | 1.27 (1.085) | 1.57 (1.174) | 1.16 (1.125) | 1.88 (0.854)
  5 minutes post challenge | 1.34 (1.068) | 1.40 (1.108) | 1.23 (1.109) | 2.12 (0.854)
  3 minutes post challenge | 0.92 (0.989) | 1.01 (0.931) | 0.86 (0.889) | 2.06 (0.912)

2. Secondary Outcome: Ciliary Redness Evaluated by the Investigator
Description: Ciliary redness and episcleral redness were evaluated by the investigator at 7, 15, and 20 minutes post-CAC using a 4-point (0 indicating none and 4 indicating extremely severe i.e. large, numerous, dilated blood vessels characterized by unusually severe deep red color, regardless of grade of chemosis, which involves the entire vessel bed) scale with half-unit (1-step) increments allowed.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1334 H 0.15% | 1334 H-0.3% | 1334 H-0.45% | Vehicle
Number analyzed (Participants) | 30 | 26 | 29 | 29
units on a scale
  20 minutes post challenge | 0.75 (0.504) | 1.05 (0.700) | 0.88 (0.553) | 1.04 (0.571)
  15 minutes post challenge | 0.70 (0.433) | 0.99 (0.740) | 0.73 (0.472) | 0.92 (0.543)
  7 minutes post challenge | 0.34 (0.344) | 0.64 (0.609) | 0.50 (0.275) | 0.62 (0.446)

ADVERSE EVENTS:
Arm/Group | 1334 H 0.15% | 1334 H-0.3% | 1334 H-0.45% | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/30 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 6/31 | 6/30 | 12/31 | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1334 H 0.15% (N=31) | 1334 H-0.3% (N=30) | 1334 H-0.45% (N=31) | Vehicle (N=30)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1334 H 0.15% (N=31) | 1334 H-0.3% (N=30) | 1334 H-0.45% (N=31) | Vehicle (N=30)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
anterior chamber cell (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anterior Chamber Pigmentation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid Exfoliation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign Body Sensation in Eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (3) | 7 (7) | 8 (8)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid Oedema (Eye disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Of the total of 122 subjects, 8 subjects did not complete the study: 114 subjects completed the study, PP population, comprised of all subjects who completed the study with no protocol violations, totaled 107 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other